CLINICAL TRIAL: NCT02614859
Title: Bicalutamide With or Without Metformin for Biochemical Recurrence in Overweight or Obese Prostate Cancer Patients (BIMET-1)
Brief Title: Bicalutamide With or Without Metformin for Biochemical Recurrence in Overweight or Obese Prostate Cancer Patients
Acronym: BIMET-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU-079; 15-1015 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation; bicalutamide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation and Bicalutamide (Active Comparator): Cycles 1-2: Observation without treatment Cycles 3-8: Bicalutamide 50 mg daily continuously to end of study
  Interventions: Drug: Observation and Bicalutamide
- Metformin and Bicalutamide (Experimental): Cycles 1-2: Metformin 1000mg BID Cycles 3-8: Bicalutamide 50 mg daily and Metformin 1000 mg BID
  Interventions: Drug: Metformin and Bicalutamide

INTERVENTIONS:
Drug: Observation and Bicalutamide — Cycles 1 - 2: Observation without treatment Cycles 3 - 8: Bicalutamide 50 mg daily, orally, continuously to the end of study (week 32).
  Arms: Observation and Bicalutamide
Drug: Metformin and Bicalutamide — Cycles 1-2: Metformin 1000mg BID Cycles 3-8: Bicalutamide 50 mg daily and Metformin 1000 mg BID
  Arms: Metformin and Bicalutamide

SUMMARY:
Obesity and metabolic syndrome are prevalent among prostate cancer patients. Having an elevated insulin level in the blood is associated with a shorter median time to cancer progression and median overall survival in patients with an elevated PSA after prior treatment. Androgen deprivation therapy (ADT) with drugs like bicalutamide is frequently used in this patient population,with no proven benefit, which may increase mortality and morbidity.This study evaluates how metformin in combination with bicalutamide affects prostate cancer.

DETAILED DESCRIPTION:
1 Cycle = 28 days = 4 weeks. Treatment will be administered on an outpatient basis ӿ Metformin starting dose is 500 mg BID, will be gradually increased to target dose of 1000mg BID.

Treatment ARM A Cycles 1 - 2: Observation without treatment Cycles 3 - 8: Bicalutamide 50 mg daily, orally, continuously to the end of study (week 32).

Treatment ARM B Cycles 1 - 2: In order to minimize gastrointestinal discomfort, metformin dosing will be ramped up over a period of 2 weeks. Metformin treatment will be started at 500 mg BID (Dose Level -2) and increased by an increment of 500 mg daily every week +/- 2 days provided no grade 2 or higher gastrointestinal toxicity is noted. If grade 2 or greater gastrointestinal toxicity occurs during the first 4 weeks of treatment, the subject will be evaluated every 2 weeks until resolution of toxicity to grade 0 or 1 and, then, the metformin dose will be increased to the next dose level. The target dose of metformin is 1000 mg BID.

ELIGIBILITY:
Inclusion Criteria:

Ability to understand and the willingness to sign a written informed consent

Male 18 years or older

Histologically or cytologically confirmed diagnosis of prostate cancer

Patient must have had previous treatment with definitive surgery or radiation therapy or cryoablation

Patient may have prior salvage therapy (surgery, radiation or other local ablative procedures) within 6 months prior to randomization if the intent was for cure.Prophylactic radiotherapy to prevent gynecomastia within 4 weeks prior to randomization is allowed BMI > 25 at study entry

Patient may have had prior neoadjuvant and/or adjuvant therapy (chemotherapy, vaccines or experimental agents) within 4 weeks prior to randomization, if the PSA rise and PSADT were documented after the testosterone level was > 150ng/dL.

Patient must have hormone-sensitive prostate cancer as evident by a serum total testosterone level > 150 ng/dL within 12 weeks prior to randomization.

PSA must be < 30 ng/mL at study entry

Patient may not have had therapy modulating testosterone levels (such as luteinizing hormone,releasing-hormone agonists/antagonists and antiandrogens) within 1 year prior to randomization, unless it was in the neoadjuvant and/or adjuvant setting

Patient must have evidence of biochemical failure after primary therapy and subsequent progression. Biochemical failure is declared when the PSA reaches a threshold value after primary treatment and it differs for radical prostatectomy or radiation therapy.

1. For radical prostatectomy the threshold for this study is PSA ≥ 0.2ng/mL
2. For radiation therapy the threshold is a PSA rise of 2 ng/mL above the nadir PSA achieved post radiation with or without hormone therapy (2006 RTOG-ASTRO Consensus definition).
3. PSA progression requires a PSA rise above the threshold measured at any time point since the threshold was reached.

PSA doubling time between 3 and 9 months. PSA calculation requires two consecutive PSA rises (PSA2 and PSA3) above the threshold PSA (total 3 PSA values); PSA2 and PSA3 must be obtained within 12 months of study entry. All baseline PSAs should be obtained at the same reference lab. Patient's PSA doubling time must be calculated using the following formula (http://www.mskcc.org/nomograms/prostate/psa doubling-time):

ECOG performance status less than or equal to 2

Ability to swallow the study drugs

Subjects must have normal organ and marrow function as defined below:

1. Absolute neutrophil count greater than or equal to 1,000/mL
2. Hemoglobin greater than or equal to 10 g/dL
3. Platelets greater than or equal to 100,000/mL
4. Total bilirubin within normal institutional limits
5. AST(SGOT)/ALT(SGPT) less than or equal to 1.5 X institutional ULN
6. Creatinine clearance greater than or equal to 60 mL/min/1.73 m2
7. Hgb A1c ≤ 6.5

Exclusion Criteria:

Evidence of metastatic disease on imaging studies (CT and/or bone scan)

Diagnosis of diabetes mellitus defined as

1. Fasting blood glucose > 126 mg/dl or,
2. Random blood glucose > 200 mg/dl
3. Hemoglobin A1C > 6.5%

Need for treatment with any conventional modality for prostate cancer (surgery, radiation therapy, and hormonal therapy)

Prior hormonal therapy for recurrent prostate cancer (hormonal therapy given in a neoadjuvant or adjuvant setting and greater than 6 months before entry is acceptable)

Treatment within the last 30 days with any investigational drug

Radiation therapy within prior 6 months (prophylactic radiotherapy to prevent gynecomastia within 4 weeks prior to randomization is allowed)

Known hypersensitivity to metformin

Prior history of lactic acidosis

Any history of myocardial infarction in the past 12 months

Subjects who consume more than 3 alcoholic beverages per day Subjects with serious intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other nonmalignant medical or psychiatric illness that is uncontrolled or whose control may be jeopardized by the complications of this therapy or may limit compliance with the study requirements (at the discretion of the investigator)

Patient with previous or concurrent malignancy. Exceptions are made for patients who meet any of the following conditions: Basal cell or squamous cell carcinoma of the skin or prior malignancy that has been adequately treated and patient has been continuously disease free for ≥ 2 years.

Subjects currently treated with metformin and/or bicalutamide or who have been treated with metformin and/or bicalutamide in the past 6 months.

Subjects who have taken 5a-reductase inhibitors (finasteride or dutasteride), saw palmetto, or PC-SPES within the last 6 weeks are ineligible. Subjects will be eligible for the study after the wash out period of 6 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Geynisman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - National Cancer Institute, Bethesda, Maryland
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bilusic M, Toney NJ, Donahue RN, Wroblewski S, Zibelman M, Ghatalia P, Ross EA, Karzai F, Madan RA, Dahut WL, Gulley JL, Schlom J, Plimack ER, Geynisman DM. A randomized phase 2 study of bicalutamide with or without metformin for biochemical recurrence in overweight or obese prostate cancer patients (BIMET-1). Prostate Cancer Prostatic Dis. 2022 Apr;25(4):735-740. doi: 10.1038/s41391-022-00492-y. Epub 2022 Jan 25. PMID 35079115

RESULTS

PARTICIPANT FLOW:
Groups:
- Bicalutamide: Bicalutamide 50 mg daily beginning at cycle 3 to cycle 8
- Metformin and Bicalutamide: Metformin 1000mg twice a day Bicalutamide 50 mg daily beginning at cycle 3
Period: Overall Study
Arm/Group | Bicalutamide | Metformin and Bicalutamide
Started | 9 | 20
Completed | 9 | 19
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participant in metformin and bicalutamide arm removed from study due to non-compliance
Groups:
- Total: Total of all reporting groups
Arm/Group | Bicalutamide | Metformin and Bicalutamide | Total
Number analyzed (Participants) | 9 | 20 | 29
Age, Continuous [Mean (Full Range); unit: years] | 63 [54 to 68] | 64 [53 to 75] | 63.7 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 20 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 6 | 19 | 25
  Black or African American | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 20 | 29

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response Rate Based on PSA
Description: Participants with undetectable PSA after 32 weeks
Time Frame: 32 weeks
Population: 29 patients were found eligible and randomized, 28 patients completed all 32 weeks of the trial, and one patient in Arm B was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide | Metformin and Bicalutamide
Number analyzed (Participants) | 9 | 19
Participants | 3 | 5

2. Secondary Outcome: PSA Decline ≥ 85% at 32 Weeks
Description: Number of patients with PSA decline ≥ 85% after 32 weeks
Time Frame: 32 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Cycles 1-2: Observation without treatment Cycles 3-8: Bicalutamide 50 mg daily continuously to end of study
  Bicalutamide: Cycles 1 - 2: Observation without treatment Cycles 3 - 8: Bicalutamide 50 mg daily, orally, continuously to the end of study (week 32).
- Arm B: Cycles 1-2: Metformin 1000mg BID Cycles 3-8: Bicalutamide 50 mg daily and Metformin 1000 mg BID
  Metformin and Bicalutamide: Cycles 1-2: Metformin 1000mg BID Cycles 3-8: Bicalutamide 50 mg daily and Metformin 1000 mg BID
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 9 | 19
Participants | 6 | 10

3. Secondary Outcome: PSA Decline
Description: Number of patients with PSA decline after 8 weeks (observation vs metformin)
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide | Metformin and Bicalutamide
Number analyzed (Participants) | 9 | 19
Participants | 1 | 8

4. Secondary Outcome: Median PSA Decline
Description: Median PSA decline after 8 weeks % (range)
Time Frame: 8 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Bicalutamide | Metformin and Bicalutamide
Number analyzed (Participants) | 9 | 19
percent change | NA [0 to 0] — Only 1 patient had a PSA decline in Arm A | 9 [4 to 24]

5. Secondary Outcome: BMI Decline After 32 Weeks
Description: Number of patients with BMI decline after 32 weeks
Time Frame: 32 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 9 | 19
Participants | 4 | 12

ADVERSE EVENTS:
Time Frame: 4 years 1 month
Description: Participants will be followed every 12 months (+/- 2 months) for up to 4 years 1 month from end of treatment for survival, adverse events, and disease status
Arm/Group | Bicalutamide | Metformin and Bicalutamide
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/19
Other Adverse Events (participants affected / at risk) | 9/9 | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bicalutamide (N=9) | Metformin and Bicalutamide (N=19)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 8
Gynecomastia (Reproductive system and breast disorders) | 3 | 4
Breast Pain (Reproductive system and breast disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 5
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 8
Nausea (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Bloating (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 4
Weight loss (Investigations) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 2
Investigations - Other (Investigations) | 1 | 2
Cholesterol high (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Fatigue (General disorders) | 2 | 5
General disorders and administration site conditions (General disorders) | 2 | 1
Edema limbs (General disorders) | 2 | 0
Pain (General disorders) | 1 | 1
Injection site reaction (General disorders) | 1 | 1
Hot flashes (Vascular disorders) | 3 | 3
Hypertension (Vascular disorders) | 0 | 2
Flushing (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 0 | 3
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-apular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02614859/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT02614859/ICF_001.pdf